CLINICAL TRIAL: NCT05121116
Title: Effects of Mindfulness Training on Autobiographical Memory
Brief Title: Effects of Mindfulness Training on Memories of Personal Past Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aleksandra Eriksen Isham (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Aleksandra Eriksen Isham, PhD, University of St Andrews
Organization: University of St Andrews (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StAMBSR1
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Depression; Mindfulness-Based Stress Reduction
Keywords: Depression vulnerability; Mindfulness-Based Stress Reduction; Randomised controlled trial; Waitlist control
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized waitlist-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention condition (Experimental): Participation in an 8-week, online, self-directed MBSR program.
  Interventions: Behavioral: Online Mindfulness-Based Stress Reduction (MBSR)
- Waitlist control condition (No Intervention): Participants in the waitlist control condition received no active intervention during the trial period but received a link to the MBSR program after completing the post-intervention assessments.

INTERVENTIONS:
Behavioral: Online Mindfulness-Based Stress Reduction (MBSR) — Participation in an 8-week MBSR program consisting of pre-recorded mindfulness practices, including a guided body scan in week 1, guided sitting meditation in week 2, mindful yoga practices in week 3 and 4, meditation on difficult emotions in week 5, visualization meditation in week 6, lovingkindness meditation in week 7, and a silent meditation in week 8. Most practices last approximately 30 minutes and participants were encouraged to engage in a mindfulness practice daily or as often as possible. In weeks 2 - 8 participants could choose to alternate the practice introduced each week with practices from previous weeks. Participants had immediate access to all practices but were asked to complete them sequentially and in the order described above over a period of eight weeks. The MBSR program also encourages participants to employ mindfulness in their daily lives, and gives access to educative readings and videos related to the weekly mindfulness practices.
  Arms: Active intervention condition

SUMMARY:
The purpose of the study was to assess the effects of participation in an online Mindfulness-Based Stress Reduction (MBSR) program on everyday memories of personal past events in individuals with depression vulnerability. Previous research has demonstrated that individuals with depression experience various difficulties when thinking about personal past events, such as more intense negative emotions, difficulties in regulating their emotions, and difficulties in recalling highly contextualized and detailed events. Some of these difficulties may continue following recovery from depression and as such may constitute a vulnerability for recurring depression. Other studies have found that mindfulness-based interventions (MBIs) may influence how people experience and regulate their emotions, and certain aspects of how people remember personal past events. Therefore, it is possible that MBIs may also influence how individuals with depression vulnerability emotionally process memories of personal past events. In the present study participants with a history of depression were allocated to either an 8-week online MBSR condition where participants were introduced to and engaged in different mindfulness practices, or a waitlist-control condition, where participants did not receive any active training or treatment. In order to assess the effects of the MBSR program on everyday memories of personal past events participants were asked to complete a memory diary in which participants recorded both spontaneously arising and word-cued memories of personal past events in everyday life, before and after participating in the MBSR program or the waitlist-control condition. The investigators hypothesized that participants in the MBSR condition would report reduced difficulties related to memories of personal past events compared to the waitlist-control group, including how participants emotionally process these memories. The investigators predicted that these effects would be greater for spontaneously occurring memories than for voluntary memories, since previous research comparing individuals with different levels of mindfulness skills suggests that mindfulness may be especially beneficial for influencing emotion regulation in response to memories that come to mind spontaneously.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effects of an online, self-directed Mindfulness-Based Stress Reduction (MBSR) program on emotion regulation in response to everyday involuntary and voluntary (word-cued) autobiographical memories in individuals with a history of depression

SECONDARY AND EXPLORATORY OBJECTIVES:

I. Determine whether an online, self-directed MBSR program performs similar to MBIs in previous studies in terms of effects on depression symptoms, trait mindfulness, and trait emotion regulation; and whether the effects of this program are similar for trait and state measures of emotion regulation.

II. Determine the effects of an online, self-directed MBSR program on additional aspects of involuntary and voluntary autobiographical memories in individuals with a history of depression, including memory specificity, centrality, and emotional experience in response to the memories.

PARTICIPANT RECRUITMENT:

Participant recruitment was done as part of a larger research project on mindfulness and autobiographical memory in depression vulnerability, which recruited both individuals with and without a depression history. The outlined study uses data from a sample of remitted depressed participants.

STUDY OUTLINE:

Participants were randomly allocated to either an 8-week active MBSR condition, or a waitlist-control condition. Participants in both conditions received information about mental health support organizations and student support options on campus following enrollment in the study.

Participants assigned to the active MBSR intervention participated in an 8-week, self-directed MBSR program which is freely available online (www.palousemindfulness.com). This MBSR program consists of a guided body scan in week 1, guided sitting meditation in week 2, mindful yoga practices in week 3 and 4, meditation on difficult emotions in week 5, visualization meditation in week 6, lovingkindness meditation in week 7, and a silent meditation in week 8. Most mindfulness practices are planned to last approximately 30 minutes and participants are encouraged to engage in a mindfulness practice daily or as often as possible. In weeks 2 - 8 participants could choose to alternate the practice introduced each week with practices from previous weeks. In addition to the formal mindfulness practices described above, the MBSR program encourages participants to employ mindfulness in their daily lives and gives access to educative readings and videos related to the weekly mindfulness practices. Participants in the active intervention had immediate access to all MBSR practices on the website but were asked to complete the practices sequentially and in the order described above over a period of eight weeks.

Participants in the waitlist-control condition did not receive any intervention during the trial, but were given a link to the MBSR program after completing the study.

In order to determine the effects of the MBSR program on everyday autobiographical memories, all participants recorded everyday involuntary and voluntary (word-cued) autobiographical memories in a naturalistic memory diary, and rated the memories along several dimensions, including emotion regulation, emotional experience, memory specificity, and centrality. Participants also completed self-report measures of depression symptoms, trait mindfulness, trait emotion regulation, personal past events, and intervention adherence.

HYPOTHESES PRIMARY OBJECTIVE:

I. The investigators hypothesized that participants in the MBSR condition would show decreased memory suppression, expressive suppression, brooding, and reflection, and increased cognitive reappraisal and non-reactivity in response to autobiographical memories compared to the waitlist-control group. The investigators predicted that these effects would be greater for involuntary than for voluntary memories, since previous research on trait mindfulness and emotion regulation in response to autobiographical memories suggests that mindfulness skills may be especially beneficial for influencing emotion regulation in response to memories that come to mind involuntarily.

ELIGIBILITY:
Inclusion Criteria:

* Native or fluent English speaker
* Being 18-65 years old
* At least one past major depressive episode

Exclusion Criteria:

* Current depressive episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Change in the employment of emotion regulation strategies in response to everyday involuntary and voluntary autobiographical memories from baseline to post-intervention | Baseline to post-intervention, an average of 11 weeks
  Self-rated (1 = Not at all, to 5 = A great deal) memory suppression ("I tried not to keep thinking about it"), expressive suppression ("I controlled my emotion by not expressing it"), reflection ("I analyzed the event to try to understand my feelings"), brooding ("I thought: Why do I always react this way?", cognitive reappraisal ("I changed the way I was thinking about the situation"), and non-reactivity ("I noticed the memory and feelings without having to react to them") in response to autobiographical memories was measured with a naturalistic memory diary method. Participants were asked to record and rate involuntary autobiographical memories in the memory diary immediately upon retrieval, over a period of up to five days or until they had recorded seven memories. For each involuntary memory recorded in the memory diary, participants were instructed to record and rate a word-cued (voluntary) memory when they had time later that day.

SECONDARY OUTCOMES:
Change in depression symptoms from baseline to post-intervention | Baseline through study completion, an average of 11 weeks
  Self-report measure: Depression, Anxiety, Stress Scales (DASS)
Change in trait mindfulness from baseline to post-intervention | Baseline to post-intervention, an average of 11 weeks
  Self-report measure: Five Facet Mindfulness Questionnaire (FFMQ)
Change in thought suppression from baseline to post-intervention | Baseline to post-intervention, an average of 11 weeks
  Self-report measure: White Bear Suppression Inventory (WBSI)
Change in expressive suppression and cognitive reappraisal from baseline to post-intervention | Baseline to post-intervention, an average of 11 weeks
  Self-report measure: Emotion Regulation Questionnaire (ERQ)
Change in rumination (brooding, reflection, overall) from baseline to post-intervention | Baseline to post-intervention, an average of 11 weeks
  Self-report measure: Ruminative Response Scale (RRS)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Dritschel, Principal Investigator — University of St Andrews
Locations (1):
- University of St Andrews, St Andrews, Ingen Region, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The raw data underpinning this study cannot be made available to other researchers due to ethical concerns since there is not agreement from the participants to share their data.

REFERENCES:
- [Background] Isham AE, del Palacio-Gonzalez A, Dritschel B. Trait Mindfulness and Emotion Regulation upon Autobiographical Memory Retrieval during Depression Remission. Mindfulness. 2020;11(12):2828-40.